CLINICAL TRIAL: NCT00268788
Title: A Controlled Cross-Over Trial of Subcutaneous Versus Intravenous Immunoglobulin for Multifocal Motor Neuropathy
Brief Title: Subcutaneous Immunoglobulin Treatment for Multifocal Motor Neuropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Thomas Harbo, Aarhus University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2005-130; EudraCT-number: 2005-000934-19
Record Dates: First submitted 2005-12-21; First posted 2005-12-22 (Estimated); Last update posted 2008-02-21 (Estimated); Status verified 2008-02

CONDITIONS: Multifocal Motor Neuropathy
Keywords: multifocal motor neuropathy; subcutaneous; IVIG; gammaglobulin
MeSH Terms: interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Subcutaneous Ig given twice a week.
  Interventions: Drug: Subcutaneous immunoglobulin
- 2 (Active Comparator): Intravenous Ig
  Interventions: Drug: Intravenous immunoglobulin

INTERVENTIONS:
Drug: Subcutaneous immunoglobulin — Individually dosed, given twice a week.
  Other Names: Subcuvia
  Arms: 1
Drug: Intravenous immunoglobulin — Individual dose and frequency
  Other Names: Endobulin
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the effect of subcutaneous administration of immunoglobulin compared to intravenous treatment, for multifocal motor neuropathy

NB. ONLY RECRUITING FROM DENMARK

DETAILED DESCRIPTION:
Introduction Intravenous immunoglobulin (IVIG) treatment is the only established treatment modality in Multifocal Motor Neuropathy (MMN). In order to maintain neuromuscular performance patients require lifelong treatment. Hospital-based treatments have high cost and inconveniences to patients, particularly in chronic disorders. Immunoglobulin preparations are now available for subcutaneous use as IgG replacement therapy. The safety and efficacy of subcutaneous infusion is reported to be comparable to i.v. preparations, and has been applied successfully in other autoimmune disorders. However patients with MMN have not previously been treated with subcutaneous immunoglobulin.

Hypothesis:

Subcutaneous immunoglobulin treatment is efficacious and safe with less patient inconvenience.

Primary endpoint:

Isokinetic muscle strength at the end of treatment A vs B (subcutaneous vs i.v.)

Secondary endpoint:

Medical research council score (MRC-score), 9-hole peg test, 10m walking, Nerve conduction parameters, SF-36.

ELIGIBILITY:
Inclusion Criteria:

- Clinical diagnosis of multifocal motor neuropathy, supported by electrophysiological findings

Exclusion Criteria:

* Other severe medical conditions
* Pregnancy and lactation
* Anti-coagulation therapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2005-08; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Isokinetic muscle strength at the three most affected muscle groups. | At the end of each arm of the crossover study

SECONDARY OUTCOMES:
Medical research council score (MRC-score), | At the end of each treatment arm of the crossover study
9-hole peg test, | At the end of each treatment arm of the crossover study
10m walking, | At the end of each treatment arm of the crossover study
Nerve conduction parameters, | At the end of each treatment arm of the crossover study
SF-36 | At the end of each treatment arm of the crossover study
Adverse effects | During each treatment arm of the crossover study

CONTACTS AND LOCATIONS:
Overall Officials: Henning Andersen, MD, DMSc, Principal Investigator — Aarhus University Hospital; Johannes Jakobsen, Professor, Study Chair — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Department of Neyrology, Aarhus, Denmark

REFERENCES:
- [Derived] Harbo T, Andersen H, Hess A, Hansen K, Sindrup SH, Jakobsen J. Subcutaneous versus intravenous immunoglobulin in multifocal motor neuropathy: a randomized, single-blinded cross-over trial. Eur J Neurol. 2009 May;16(5):631-8. doi: 10.1111/j.1468-1331.2009.02568.x. Epub 2009 Feb 19. PMID 19236457